CLINICAL TRIAL: NCT03462875
Title: The ENIGMA Study: Eastern Inflammatory Bowel Disease Gut Microbiota
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Melbourne (Other); The University of Queensland (Other); Sun Yat-sen University (Other); Kunming Medical University (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: ENIGMA II
Record Dates: First submitted 2018-02-12; First posted 2018-03-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Dietary pattern; Environmental factors; Gut microbiota
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Crohn's Disease Patients: Subjects having confirmed diagnosis of Crohn's disease which is defined by endoscopy, radiology and histology; and having documented ileocaecal or right-sided colonic disease
- Non-household Controls: Non-affected subjects who will under colonoscopy for polyp or colorectal cancer screening, or investigations of gastrointestinal symptoms other than Inflammatory Bowel Disease
- First Degree Relatives: Non-affected first degree relatives of cases
- Household/co-habitant Controls: Non-affected subjects living in the same household with the cases in the recent 6 months

SUMMARY:
The incidence of inflammatory bowel diseases, (IBD) including Crohn's disease (CD) and ulcerative colitis (UC), is increasing in the developing world. Our recent Asia-Pacific population-based study in 8 Asian countries and Australia has demonstrated that Hong Kong and China have amongst the highest disease incidences in Asia while Australia has the equal highest incidence of these diseases in the world.

The ENIGMA project comprises three main enteric microbiome domains of central importance to Crohn's disease. Two specific organisms which may play a critical role in disease pathogenesis, including the candidate protective bacterium, and the novel pathogenic candidate, will be characterized and studied in detail. Microbial findings will be related to a detailed assessment of environmental factors that permit microbial changes or expression.

DETAILED DESCRIPTION:
The incidence of inflammatory bowel diseases, (IBD) including Crohn's disease (CD) and ulcerative colitis (UC), is increasing in the developing world. Our recent Asia-Pacific population-based study in 8 Asian countries and Australia have demonstrated that Hong Kong and China have amongst the highest disease incidences in Asia while Australia has the equal highest incidence of these diseases in the world. The incidence of IBD in Hong Kong and China has risen three-fold in the past decade.

Asian populations have genetic predispositions to develop IBD which are different to the West, but these genetic abnormalities are not obligatory for the development of IBD, with environmental factors playing a much more important pathogenic role. These factors include travel with exposure to a new population in childhood, diet, antibiotic use during childhood, socioeconomic status, and a rural versus urban upbringing, each of which alone, or in combination, are likely to affect the microbiome.

Compelling evidence suggests that gut microbes play a critical role in disease pathogenesis, while geographic, dietary and ethnic factors impact the microbial composition. In addition to broad changes in the microbial profile in IBD, a number of specific changes have been identified, such as a decrease of the butyrate-producing species Roseburia hominis and Faecalibacterium Prausnitzii. Although the commensal gut microbiota is ecologically and functionally perturbed in IBD, there is unexplained heterogeneity among IBD subtypes and individual patients. In new-onset treatment naïve patients with CD, enrichment for the Enterobacteriaceae and depletion of Clades IV and XIVa Clostridia during disease-associated inflammation have been reported. Metagenomic studies and microarray analyses in Western populations and limited Asian data have demonstrated a reduction of Firmicutes, such as F. prausnitzii in Crohn's disease (CD), and an increased in Escherichia coli and Fusobacterium. It is unknown if the changes in putative pathogens and/or protective organisms identified in Western populations, such as E. coli and F. prausnitzii, respectively, are present in IBD patients in Asia. Information is also lacking about the degree of genetic variation between the bacteria assigned to these taxonomic groups from different ethnic and geographical regions. Most of the published work on these bacteria, and their potential pathogenic or protective role in CD, has been undertaken with isolates recovered from European and North American subjects. For these reasons, The investigators believe there is a need to firmly establish whether the microbial changes outlined above are also encountered in patients from other parts of the world, including Asian countries with high disease incidence and increasing disease incidence.

The Post-Operative Crohn's Endoscopic Recurrence (POCER) study was undertaken in 17 hospitals around Australia and New Zealand and recruited 174 patients who were then monitored for 18 months post-operatively. The microbiota analyses undertaken on a subset of the POCER study patient cohort showed that F. prausnitzii, previously identified as being capable of producing anti-inflammatory properties possible key organism in preventing active CD were decreased in abundance in active CD, in patients at the surgery who subsequently recurred, and in patients at the time of recurrence. Most of the published studies examining the anti-inflammatory properties of F. prausnitzii have been undertaken with a single strain of European origin. Despite the promise associated with the anti-inflammatory properties produced by F. prausnitzii it remains to be determined whether this bacterium is protective against inflammation, or diminishes subsequent to the onset of inflammation.

In summary, it is currently unclear if the changes in putative pathogens and protective organisms present in Western IBD populations are consistently observed with CD patients in Asia. Nor is it known whether the functional capabilities of these bacteria differ across ethnic and/or geographic regions.

In addition to the characteristics of these two bacterial families, the microbial environment interfacing with these organisms is likely to play a critical role in their expression and function. This will be examined in detail using broad sequencing techniques.

Microbial analyses will be undertaken in the context of a detailed examination of environmental risk factors for the development of CD, in the same patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years old
2. competent to provide informed consent (no mental illness or dementia, etc. that will hinder the understanding)
3. living in the same area for recent 6 months

Exclusion Criteria:

1. Use of anticoagulants within 1 week
2. Use of prebiotics, probiotics or antibiotics in recent 3 months
3. Use of laxatives or "Stoppers" in the last 3 months
4. Vaccination within 3 months
5. Recent dietary changes (e.g. becoming vegetarian/vegan)
6. Known complex infections or sepsis (excl. simple infections such as influenza etc.)
7. Known history or concomitant significant food allergies
8. Known history of severe organ failure (including decompensated cirrhosis, malignant disease, kidney failure, epilepsy, active serious infection, acquired immunodeficiency syndrome)
9. Bowel surgery in the last 6 months (excluding colonoscopy/ procedure related to perianal disease)
10. Having stoma
11. Known pregnancy
12. Travel history within 4 weeks (need to define the travel history in China)
13. Known contraindications to colonoscopy
14. Colonoscopy in the last month prior to sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Cases are those subjects having confirmed diagnosis of Crohn's disease which is defined by endoscopy, radiology and histology; and having documented ileocaecal or right-sided colonic disease;
  2. Non-household controls are non-affected subjects who will under colonoscopy for polyp or colorectal cancer screening, or investigations of gastrointestinal symptoms other than Inflammatory Bowel Disease
  3. Household/co-habitant controls are non-affected subjects living in the same household with the cases in the recent 6 months
  4. FDR are the non-affected first degree relatives of cases.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Identification of Key Microbiota | 2 years
  To study key identified bacteria and broader aspects of the microbiota that may play a role in Crohn's disease pathophysiology, in patients and healthy controls, in Asian and Western populations

SECONDARY OUTCOMES:
Influence of Dietary Factors | 2 years
  To address the influence of dietary additives exposures on the etiology and prevalence of Inflammatory Bowel Diseases
Influence of Environmental Factors | 2 years
  To address the influence of environmental exposures on the etiology and prevalence of Inflammatory Bowel Diseases
Relationship between environmental factor and Crohn's disease | 2 years
  To evaluate which environmental factors will cause Crohn's disease
Relationship between environmental factor and Crohn's disease related Mircobiota | 2 years
  To evaluate the environmental factors and the microbiota in Crohn's disease
Target Therapy for Crohn's Disease | 2 years
  To target microbial factors as therapy in Crohn's disease

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong